CLINICAL TRIAL: NCT05076786
Title: Chidamide Plus Etoposide and Cisplatin/Carboplatin as First-line Treatment for Advanced Extrapulmonary Neuroendocrine Carcinoma: a Prospective, Multicenter, Single-arm, Phase 2 Clinical Study
Brief Title: Chidamide Plus Etoposide and Cisplatin/Carboplatin as First-line Treatment for Extrapulmonary Neuroendocrine Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The First Affiliated Hospital of Xiamen University (Other); Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-3125
Record Dates: First submitted 2021-09-18; First posted 2021-10-13 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-09

CONDITIONS: Neuroendocrine Tumors; Neuroendocrine Carcinoma
Keywords: Histone Deacetylase Inhibitors; Chidamide; Neuroendocrine Carcinoma
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Etoposide; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide + Etoposide + Cisplatin/Carboplatin (Experimental): Experimental arm will be treated by chidamide combined with etoposide and cisplatin/carboplatin regimen for 4-6 cycles.
  Interventions: Drug: Chidamide; Drug: Etoposide + Cisplatin/Carboplatin

INTERVENTIONS:
Drug: Chidamide — 20mg, administered orally. Week 1/2: twice a week (d0, d4, d7, d11); Week 3: stop. Repeat every 3 weeks for 4-6 cycles.
  Other Names: Epidaza
Drug: Etoposide + Cisplatin/Carboplatin — Etoposide (100mg/m2; intravenous infusion; d1-3) + Cisplatin (75mg/m2; intravenous infusion; d1). Repeat every 3 weeks for 4-6 cycles.
  OR Etoposide (100mg/m2; intravenous infusion; d1-3) + Cisplatin (25mg/m2; intravenous infusion; d1-3). Repeat every 3 weeks for 4-6 cycles.
  OR Etoposide (100mg/m2; intravenous infusion; d1-3) + Carboplatin (AUC=5; intravenous infusion; d1). Repeat every 3 weeks for 4-6 cycles.
  Other Names: EP/EC regimen

SUMMARY:
The purpose of this study is to explore the efficacy and safety of chidamide combined with etoposide and cisplatin/carboplatin in the first-line treatment of advanced extrapulmonary neuroendocrine carcinoma.

DETAILED DESCRIPTION:
This study is a single-arm, multi-center, two-stage, phase II clinical trial conducted in China. This study adopts Simon's two-stage design, and the inclusion criteria and exclusion criteria of the two stages were consistent. Twelve patients with extrapulmonary neuroendocrine carcinoma will be enrolled in the first stage. If more than four complete or partial responses were seen at planned interim analysis, the additional 16 patients will be recruited in the second stage and a total of 28 patients will be treated.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Histologically confirmed locally advanced and metastatic extrapulmonary neuroendocrine carcinoma;
3. No systematic treatments for neuroendocrine carcinoma are received before enrollment;
4. ECOG ≤ 2;
5. Have at least one measurable lesion according to RECIST version 1.1, and the lesion has not received any local treatments;
6. Absolute neutrophil count ≥ 1.5×109 / L, platelet count ≥ 100×109 / L, hemoglobin ≥ 90 g/L;
7. Have ability to sign a written informed consent.

Exclusion Criteria:

1. Have surgery or trauma within 4 weeks before enrollment, or are expected to receive surgical treatment;
2. Previous use of HDAC inhibitors;
3. Allergy to related drug components;
4. Have a medical history of immune deficiency diseases, or organ transplantation;
5. Have uncontrolled or significant cardiovascular disease;
6. Abnormal liver function (total bilirubin > 1.5×upper limit of normal); Transaminases (ALT/AST) >2.5×upper limit of normal (>5x upper limit of normal for patients with liver metastases), abnormal renal function (serum creatinine > 1.5×upper limit of normal);
7. Pregnancy ;
8. Have serious diseases that may endanger the safety of patients, or affect patients to complete the research;
9. Any serious mental or cognitive disorder;
10. Patients are currently enrolled in another drug clinical trial within 4 weeks prior to enrollment;
11. Any other condition which is inappropriate for the study in the opinion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  Percentage of participants with complete response and partial response, assessed by the investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 2 years
  Percentage of participants with complete response, partial response, and stable disease assessed by the investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1
Progression-free Survival (PFS) | Time from the date of enrollment to the earliest of documented disease progression or death, assessed up to 2 years
  Time from the date of enrollment until progression or death, whichever is first met
Overall Survival (OS) | Time from the date of enrollment to the earliest of documented death, assessed up to 3 years
  Time from the date of enrollment until death
Treatment-related Adverse Events (Safety) | Up to 2 years
  Frequency and grade of adverse events (the grade of adverse events is assessed according to CTCAE v4.03).

CONTACTS AND LOCATIONS:
Overall Officials: Chunmei Bai, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (3):
- China (3):
  - Department of Medical Oncology, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not available to others.